CLINICAL TRIAL: NCT02397577
Title: Normal Values for Gastric Emptying in a 13C-octanoate Breath Test Using a Solid Test Meal
Brief Title: Reference Values for Gastric Emptying
Acronym: 13C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-NR. 2013-0338
Record Dates: First submitted 2015-03-18; First posted 2015-03-25 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Delayed Gastric Emptying
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gastric emptying measurements (Other)
  Interventions: Other: Solid test meal, liquid test meal on two separate occations

INTERVENTIONS:
Other: Solid test meal, liquid test meal on two separate occations — 13C labeld solid test meal, 13C labeld liquid test meal on two separate occations

SUMMARY:
Healthy volunteers will ingest a 13C-octaoate containing test meal and 13C in expiratory air will be followed. Normal values will be calculated data of these tests.

DETAILED DESCRIPTION:
This is a clinical study for establishing reference values in a 13C-octanoate breath test and a 13C-sodium acetate breath test. Healthy volunteers (n=75) will eat a solid test meal of scrambled eggs and toast containing 13C-octanoate. 13C-content of exhaled air will be measured at baseline and followed for the next 4 hours. One week later, the healthy volunteers (n=75) will drink a standardized nutritional shake (Ensure Plus Vanille, Abbott) containing 13C-sodium acetate. 13C-content of exhaled air will be measured at baseline and for the next 4 hours. Estimated gastric emptying time will be calculated using established algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects free of relevant abdominal complaints
* Written informed consent

Exclusion Criteria:

* Age under 18
* Previous history of gastrointestinal disease or surgery (excludes appendectomy, hernia repair and anorectal disorders)
* Known diabetes mellitus, scleroderma, neurological impairment or other major current disease
* Subjects unable to stop medication that alters gut function for 1 week prior to the study, including anticholinergics, calcium canal inhibitors, beta blocker, prokinetics, proton-pump inhibitors, DDV-IV-Inhibitors, Inkretin-mimetica, non-steroidal anti-inflammatory drugs, macrolid antibiotics
* Pregnancy beyond week 12 (no pregnancy test will be performed)
* Involvement in any other clinical trial during the course of this trial, nor within a period of 14 days prior to its beginning or 14 days after its completion
* Known allergy or intolerance against hen egg protein or gluten

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Half gastric emptying time t50 according to Ghoos et al. (t50_Ghoos) | 4 hours after test meal

SECONDARY OUTCOMES:
t50 according to Bluck & Coward (t50_Bluck) | 4 hours after test meal
t50 according to Wagner & Nelson (t50_WN) | 4 hours after test meal
Gastric emptying coefficient (GEC) | 4 hours after test meal

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, University Hospital Zurich, Zurich, Switzerland